CLINICAL TRIAL: NCT06457204
Title: Bioequivalence of Two Sifrol® Tablets Following Oral Administration in Healthy Subjects (an Open-label, Randomised, Single-dose, Two-way Crossover Trial)
Brief Title: A Study in Healthy People to Compare Two Different Sifrol® Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0248-0689; 2024-510764-23-00 (Registry Identifier: CTIS); U1111-1303-3852 (Registry Identifier: WHO Registry (ICTRP))
Record Dates: First submitted 2024-06-10; First posted 2024-06-13 (Actual); Results first posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reference - Test (Experimental): Subjects received the reference product followed by the test product, the treatments were separated by a wash-out phase of at least 3 days.
  Reference product: Healthy subjects received 1 tablet Sifrol® (pramipexole) manufactured in Ingelheim containing 0.088 mg pramipexole taken orally after an overnight fast of at least 10 hours.
  Test product: Healthy subjects received 1 tablet Sifrol® (pramipexole) manufactured in Ennigerloh containing 0.088 mg pramipexole taken orally after an overnight fast of at least 10 hours.
  Interventions: Drug: Pramipexole manufactured in Ingelheim; Drug: Pramipexole manufactured in Ennigerloh
- Test - Reference (Experimental): Subjects received the test product followed by the reference product, the treatments were separated by a wash-out phase of at least 3 days.
  Test product: Healthy subjects received 1 tablet Sifrol® (pramipexole) manufactured in Ennigerloh containing 0.088 mg pramipexole taken orally after an overnight fast of at least 10 hours.
  Reference product: Healthy subjects received 1 tablet Sifrol® (pramipexole) manufactured in Ingelheim containing 0.088 mg pramipexole taken orally after an overnight fast of at least 10 hours.
  Interventions: Drug: Pramipexole manufactured in Ingelheim; Drug: Pramipexole manufactured in Ennigerloh

INTERVENTIONS:
Drug: Pramipexole manufactured in Ingelheim — 1 tablet Sifrol® (pramipexole) manufactured in Ingelheim containing 0.088 mg pramipexole taken orally after an overnight fast of at least 10 hours.
  Other Names: Sifrol® Tabletten
Drug: Pramipexole manufactured in Ennigerloh — 1 tablet Sifrol® (pramipexole) manufactured in Ennigerloh containing 0.088 mg pramipexole taken orally after an overnight fast of at least 10 hours.
  Other Names: Sifrol® Tabletten

SUMMARY:
The main objective of this trial is to establish the bioequivalence of Sifrol® tablets manufactured at two different sites.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female subjects according to the assessment of the investigator, as based on a complete medical histo1y including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), and clinical laboratory tests
2. Age of 18 to 55 years (inclusive)
3. Body mass index (BMI) of 18.5 to 29.9 kg/m² (inclusive)
4. Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to admission to the trial Further inclusion criteria apply.

Exclusion Criteria:

1. Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
2. Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 90 beats per minute (bpm)
3. Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
4. Any evidence of a concomitant disease assessed as clinically relevant by the investigator Further exclusion criteria apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2024-07-02 (Actual); Primary Completion 2024-08-12 (Actual); Study Completion 2024-08-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Humanpharmakologisches Zentrum Biberach, Biberach, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a randomized, open-label, two-way crossover design trial.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated
Period: Period 1
Arm/Group | Reference - Test | Test - Reference
Started | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0
Period: Washout
Arm/Group | Reference - Test | Test - Reference
Started | 14 | 14
Completed | 14 | 12
Not Completed | 0 | 2
Not completed — Adverse Event | 0 | 2
Period: Period 2
Arm/Group | Reference - Test | Test - Reference
Started | 14 | 12
Completed | 14 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): All subjects who were treated with at least one dose of trial drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Reference - Test | Test - Reference | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.9 (8.9) | 40.1 (9.7) | 39.0 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 16
  Male | 5 | 7 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 14 | 14 | 28
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 13 | 14 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of Pramipexole in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: Area under the concentration-time curve of pramipexole in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz).
  Data was derived from an Analysis of variance (ANOVA) on the logarithmic scale including effects for sequence, subjects nested within sequences, period and treatment. The effect 'subjects within sequences' were considered as random, whereas the other effects were considered as fixed. CIs were calculated based on the residual error from the ANOVA and quantiles from the t-distribution. These quantities were then back-transformed to the original scale to provide the point estimate and 90% CIs for each endpoint.
Time Frame: Within 3 hours prior to drug administration and 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 34 and 48 hours following administration.
Population: Pharmacokinetic set (PKS): all subjects in the TS who provided at least one PK endpoint that was defined as primary or secondary and was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK nonevaluability.
Measure: Geometric Least Squares Mean (Standard Error); unit: hour * picogram per milliliter
Groups:
- Reference - Sifrol® (Pramipexole) Manufactured in Ingelheim: Reference product: Healthy subjects received 1 tablet Sifrol® (pramipexole) manufactured in Ingelheim containing 0.088 mg pramipexole taken orally after an overnight fast of at least 10 hours.
- Test - Sifrol® (Pramipexole) Manufactured in Ennigerloh: Test product: Healthy subjects received 1 tablet Sifrol® (pramipexole) manufactured in Ennigerloh containing 0.088 mg pramipexole taken orally after an overnight fast of at least 10 hours.
Arm/Group | Reference - Sifrol® (Pramipexole) Manufactured in Ingelheim | Test - Sifrol® (Pramipexole) Manufactured in Ennigerloh
Number analyzed (Participants) | 26 | 27
hour * picogram per milliliter | 3573 (NA) — Adjusted geometric standard error = 1.039 | 3632 (NA) — Adjusted geometric standard error = 1.039
Statistical Analysis 1: Comparison: Reference - Sifrol® (Pramipexole) Manufactured in Ingelheim vs Test - Sifrol® (Pramipexole) Manufactured in Ennigerloh; Analysis of variance (ANOVA) on the logarithmic scale included effects for sequence, subjects nested within sequences, period and treatment. The effect 'subjects within sequences' was considered as random, whereas the other effects were considered as fixed. confidence intervals (CIs) were calculated based on the residual error from the ANOVA and quantiles from the t-distribution. These quantities were then back-transformed to the original scale to provide the point estimate and 90% CIs; Test type: Other; Ratio of adjusted geometric means [%] = 101.6, 90% CI 2-sided [98.4 to 105.0] — Ratio of adjusted geometric means [%] calculated as: test/reference*100. Intra-individual geometric coefficient of variation (gCV) [%] = 6.9

2. Primary Outcome: Maximum Measured Concentration of Pramipexole in Plasma (Cmax)
Description: Maximum measured concentration of pramipexole in plasma (Cmax).
  Data was derived from an Analysis of variance (ANOVA) on the logarithmic scale including effects for sequence, subjects nested within sequences, period and treatment. The effect 'subjects within sequences' were considered as random, whereas the other effects were considered as fixed. CIs were calculated based on the residual error from the ANOVA and quantiles from the t-distribution. These quantities were then back-transformed to the original scale to provide the point estimate and 90% CIs for each endpoint.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Standard Error); unit: picogram per milliliter
Arm/Group | Reference - Sifrol® (Pramipexole) Manufactured in Ingelheim | Test - Sifrol® (Pramipexole) Manufactured in Ennigerloh
Number analyzed (Participants) | 26 | 27
picogram per milliliter | 285 (NA) — Adjusted geometric standard error = 1.037 | 280 (NA) — Adjusted geometric standard error = 1.036
Statistical Analysis 1: Comparison: Reference - Sifrol® (Pramipexole) Manufactured in Ingelheim vs Test - Sifrol® (Pramipexole) Manufactured in Ennigerloh; [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of adjusted geometric means [%] = 98.3, 90% CI 2-sided [91.6 to 105.5] — Ratio of adjusted geometric means [%] calculated as: test/reference*100. Intra-individual geometric coefficient of variation (gCV) [%] = 15.0

3. Secondary Outcome: Area Under the Concentration-time Curve of Pramipexole in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: Area under the concentration-time curve of pramipexole in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞).
  Data was derived from an Analysis of variance (ANOVA) on the logarithmic scale including effects for sequence, subjects nested within sequences, period and treatment. The effect 'subjects within sequences' were considered as random, whereas the other effects were considered as fixed. CIs were calculated based on the residual error from the ANOVA and quantiles from the t-distribution. These quantities were then back-transformed to the original scale to provide the point estimate and 90% CIs for each endpoint.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Standard Error); unit: hour * picogram per milliliter
Arm/Group | Reference - Sifrol® (Pramipexole) Manufactured in Ingelheim | Test - Sifrol® (Pramipexole) Manufactured in Ennigerloh
Number analyzed (Participants) | 26 | 27
hour * picogram per milliliter | 3730 (NA) — Adjusted geometric standard error = 1.040 | 3788 (NA) — Adjusted geometric standard error = 1.040
Statistical Analysis 1: Comparison: Reference - Sifrol® (Pramipexole) Manufactured in Ingelheim vs Test - Sifrol® (Pramipexole) Manufactured in Ennigerloh; [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of adjusted geometric means [%] = 101.6, 90% CI 2-sided [98.2 to 105.0] — Ratio of adjusted geometric means [%] calculated as: test/reference*100. Intra-individual geometric coefficient of variation (gCV) [%] = 7.1

ADVERSE EVENTS:
Time Frame: Adverse events: up to 2 days following drug intake. All-cause mortality: up to 24 days.
Description: Treated set (TS): All subjects who were treated with at least one dose of trial drug.
Arm/Group | Reference - Sifrol® (Pramipexole) Manufactured in Ingelheim | Test - Sifrol® (Pramipexole) Manufactured in Ennigerloh
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/28
Other Adverse Events (participants affected / at risk) | 7/26 | 5/28
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Reference - Sifrol® (Pramipexole) Manufactured in Ingelheim (N=26) | Test - Sifrol® (Pramipexole) Manufactured in Ennigerloh (N=28)
Nausea (Gastrointestinal disorders) | 2 | 3
Vomiting (Gastrointestinal disorders) | 0 | 3
Dizziness (Nervous system disorders) | 3 | 0
Headache (Nervous system disorders) | 6 | 5
Orthostatic intolerance (Nervous system disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2024-04-29): https://cdn.clinicaltrials.gov/large-docs/04/NCT06457204/Prot_000.pdf
  • Statistical Analysis Plan (2024-08-23): https://cdn.clinicaltrials.gov/large-docs/04/NCT06457204/SAP_001.pdf